CLINICAL TRIAL: NCT06720558
Title: A 3-week Randomized Controlled Trial on the Efficacy of a Placebo Probiotic in Rebalancing Gut Health and Fostering Physical and Emotional Well-being in Individuals With Mild Gastrointestinal Symptoms
Brief Title: Effects of a Placebo Probiotic on Gut Health and General Well-being in Individuals With Mild Gastrointestinal Symptoms
Acronym: PlaCIBO
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Catholic University of the Sacred Heart (Other)
Responsible Party: Principal Investigator, Diletta Barbiani, Junior Assistant Professor, Catholic University of the Sacred Heart
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PlaCIBO_MtBlab
Record Dates: First submitted 2024-11-27; First posted 2024-12-06 (Actual); Last update posted 2024-12-06 (Actual); Status verified 2024-12

CONDITIONS: Healthy
Keywords: Gastrointestinal Symptoms; Placebo Effect; Open-Label Placebo

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Deceptive Placebo (Experimental)
  Interventions: Other: Placebo probiotic
- Control - Open-Label PLacebo (Other): The Control Arm will not be exposed to any intervention for the first three weeks. After this time and for the following three weeks, participants will receive placebo probiotic pills in an open-label fashion: they will be honestly informed that the pills are inert placebos.
  Interventions: Other: Open-Label Placebo probiotic; Other: Control-no treatment

INTERVENTIONS:
Other: Placebo probiotic — Three-week consumption of placebo probiotic capsules passed off as being actual probiotics
  Arms: Deceptive Placebo
Other: Open-Label Placebo probiotic — Participants of the Control group will be switched to this condition after three weeks and receive placebo probiotic capsules for the following three-weeks of no intervention. Specifically, they will be honestly informed that the capsules are inert placebos.
  Arms: Control - Open-Label PLacebo
Other: Control-no treatment — For the first three weeks, the Control group will not be exposed to any intervention.
  Arms: Control - Open-Label PLacebo

SUMMARY:
The present study is aimed at exploring whether positive expectations of receiving a three-week treatment with a probiotic supplement (in fact a placebo) improve symptoms of gastrointestinal distress and promote physical and emotional well-being in healthy individuals with mild gastrointestinal symptoms. At first, a comparison is planned between (1) a classic deceptive placebo manipulation (Deceptive Placebo group, DP), and (2) a control condition (Control group, C), in which no placebo substance will be administered. After the three-week waiting list, the Control group will be invited to take the placebo probiotic pills in an "open-label" fashion (Open Label Placebo, OLP). Specifically, participants will be informed that the pills are inert placebos. An exploratory analysis will help to clarify whether the OLP paradigm leads to significant effects, based on a within-group (C- OLP) and between-group comparison (DP-OLP).

ELIGIBILITY:
Inclusion Criteria:

* Age between 20 and 65
* Individuals with mild gastrointestinal symptoms (e.g., digestive issues, acid reflux, constipation) such that normal every-day activities are not severly compromised.

Exclusion Criteria:

* Individuals with a diagnosis of functional gastrointestinal disorders (e.g., irritable bowel syndrome, ulcerative colitis, chronic inflammatory bowel diseases).
* Individuals suffering from neurodegenerative diseases and/or psychiatric conditions
* Individuals taking probiotic supplementation at the time of enrollment in the study

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-11-20 (Actual); Primary Completion 2025-04 (Estimated); Study Completion 2025-04 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in the Gastrointestinal Symptom Rating Scale (GSRS) total score at 3 weeks. | Baseline and 3 weeks

SECONDARY OUTCOMES:
Change from Baseline in the Digestion-Associated Quality Of Life Questionnaire (DQLQ) total score at 3 weeks. | Baseline and 3 weeks
Change from Baseline in Stool Form as assessed by means of the Bristol Stool Scale | Day 2/3 and day 19/20 from Baseline
  The Bristol stool scale is a diagnostic medical tool designed to classify the form of human stool into seven categories.
Change from Baseline in Fatigue Levels as assessed by means of the Multidimensional Fatigue Inventory (MFI-20) at 3 weeks. | Baseline and 3 weeks
  Items are scored 1-5, with 10 [fatigue-]positively phrased items reverse scored (items 2, 5, 9, 10, 13, 14, 16, 17, 18, 19). In the final score, high scores represent more fatigue.
Change from Baseline in Sleepiness Levels as assessed by means of the The Epworth sleepiness scale at 3 weeks. | Baseline and 3 weeks
  Final total score ranges from 0 to 24. Scores from 0 to 10 show average (normal) daytime sleepiness. A result from 11 to 24 indicates excessive (abnormal) daytime sleepiness.
Change from Baseline in Positive and Negative affect as assessed by means of the Positive and Negative Affect Schedule (PANAS) at 3 weeks. | Baseline and 3 weeks
Change from Baseline in Stress Levels as assessed by means of the Perceived Stress Scale (PSS) 3 weeks. | Baseline and 3 weeks
  The scale comprises of 10 items, with scores ranging from 0 ( = Never) to 4 ( = Very Often). Scores ranging from 0-13 would be considered low stress. Scores ranging from 14-26 would be considered moderate stress. Scores ranging from 27-40 would be considered high perceived stress.

CONTACTS AND LOCATIONS:
Locations (1):
- Catholic University of the Sacred Heart, Milan, Italy

IPD SHARING:
Plan to Share IPD: Yes